CLINICAL TRIAL: NCT06947356
Title: A Multicenter, Prospective, Open-label, Non-inferiority Randomized Controlled Study on the Efficacy of Tenofovir Alafenamide Fumarate vs. Tenofovir Disoproxil Fumarate in Preventing Mother-to-Child Transmission of Hepatitis B Virus in Pregnant Women With High Viral Loads
Brief Title: Comparison of TAF and TDF in Preventing Mother-to-Child Transmission of HBV in Pregnancies With High Viral Loads
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou 8th People's Hospital (Other)
Responsible Party: Principal Investigator, Calvin Q.Pan, Principal Investigator, Clinical Professor, Guangzhou 8th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: US-CN-P818
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAF group (Experimental): Pregnant women will start TAF treatment (25 mg tablet taken orally once daily) from 28 weeks of gestation until delivery. After that, they will be randomly assigned to two subgroups among postpartum mothers without HBV treatment indications: one subgroup will stop treatment, while the other subgroup will continue with an additional 12 weeks of TAF treatment. The mothers and their infants will be followed up at 28 weeks postpartum. Infants will receive the hepatitis B vaccine and HBIG within 12 hours after birth, as well as booster doses of the hepatitis B vaccine at 4 weeks and 24 weeks.
  Interventions: Drug: TAF group
- TDF group (Active Comparator): The mother will start receiving TDF treatment (300 mg tablet taken orally once daily) at 28 weeks of pregnancy until delivery. After that, mothers without HBV treatment indications will be randomly assigned to two subgroups: one subgroup will stop treatment, while the other subgroup will receive an additional 12 weeks of TDF treatment. Infants will be vaccinated with the hepatitis B vaccine and HBIG within 12 hours after birth, as well as receive booster doses of the hepatitis B vaccine at 4 weeks and 24 weeks.
  Interventions: Drug: TDF group

INTERVENTIONS:
Drug: TAF group — Pregnant women will start TAF treatment (25 mg tablet taken orally once daily) from 28 weeks of gestation until delivery. After that, they will be randomly assigned to two subgroups among postpartum mothers without treatment indications: one subgroup will stop treatment, while the other subgroup will continue with an additional 12 weeks of TAF treatment. The mothers and their infants will be followed up at 28 weeks postpartum. Infants will receive the hepatitis B vaccine and HBIG within 12 hours after birth, as well as booster doses of the hepatitis B vaccine at 4 weeks and 24 weeks.
  Other Names: TAF
  Arms: TAF group
Drug: TDF group — The mother will start receiving TDF treatment (300 mg tablet taken orally once daily) at 28 weeks of pregnancy until delivery. After that, mothers without treatment indications will be randomly assigned to two subgroups: one subgroup will stop treatment, while the other subgroup will receive an additional 12 weeks of TDF treatment. Infants will be vaccinated with the hepatitis B vaccine and HBIG within 12 hours after birth, as well as receive booster doses of the hepatitis B vaccine at 4 weeks and 24 weeks.
  Other Names: TDF
  Arms: TDF group

SUMMARY:
The main objective of this study is to compare the mother-to-infant transmission rates of hepatitis B between pregnant women receiving treatment with tenofovir alafenamide and those receiving treatment with tenofovir disoproxil fumarate, after administering the hepatitis B vaccine and hepatitis B immunoglobulin to their infants at birth. Investigators define the mother-to-infant transmission rate of hepatitis B as the proportion of infants who are HBsAg positive and have serum HBV DNA >20 IU/mL at 28 weeks of age among all live births in the experimental group.

Additionally, this study will also compare the incidence of congenital defects/malformations in infants born to mothers treated with tenofovir alafenamide and tenofovir disoproxil fumarate during the perinatal period to assess drug safety.

DETAILED DESCRIPTION:
see summary

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women aged between 20 and 40 years old
2. Pregnancy duration between 20 to 28 weeks (screening for eligible patients can start from the 20th week of gestation)
3. Clinically diagnosed with compensated chronic hepatitis B, HBsAg positive for more than 6 months, with clinical history, signs, and test results consistent with compensated chronic hepatitis B
4. HBsAg and HBeAg positive in maternal serum during screening
5. PCR testing shows maternal serum HBV DNA levels exceeding 200,000 IU/mL
6. Subjects voluntarily agree to undergo treatment according to the study design's drug treatment plan and all other research requirements, and patients consent to strictly avoid pregnancy within 28 weeks postpartum
7. Patients and their husbands (the biological parents of the child) understand the risks and voluntarily participate in the study. The mother must participate voluntarily and sign a written informed consent document before participating in the study.

Exclusion Criteria:

1. Creatinine clearance < 100 mL/min (calculated using the Cockcroft-Gault method based on serum creatinine and ideal body weight), or hypophosphatemia (below normal range).
2. History of adverse renal reactions induced by Adefovir or history of Adefovir resistance.
3. Meeting one of the following criteria: hemoglobin < 80 g/L, neutrophil count < 1000/μL, ALT > 5 times the upper limit of normal, total bilirubin > 20 mg/L, albumin < 25 g/L, abnormal levels of creatinine or urea nitrogen.
4. Pregnant women with a history of miscarriage, history of giving birth to a child with congenital malformations, or history of fetal infection with hepatitis B virus.
5. The biological father of the current pregnancy has chronic hepatitis B.
6. The investigator assesses that the subject has significant kidney, cardiovascular, pulmonary, or neurological diseases that affect their participation in the study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 210 (Estimated)
Dates: Start 2025-05-03 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
The mother-to-child transmission rate of HBV | 28 weeks
  Compare the difference in HBV mother-to-infant transmission rates between pregnant women receiving TAF treatment and vaccinating their infants with hepatitis B vaccine and HBIg, and those receiving TDF treatment with the same vaccination for their infants. Here, the mother-to-infant transmission rate is defined as the proportion of infants in the experimental group who have serum HBV DNA >20 IU/mL and are HBsAg positive at 28 weeks of age among all live births.

SECONDARY OUTCOMES:
Congenital defects/malformations in infants | 28 weeks
  Determine the incidence of congenital defects/malformations in infants born to mothers treated with TAF and TDF during the perinatal period, and then conduct a comparative analysis of these data.
The percentage of mothers in each group of pregnant women with HBV DNA below 200,000 IU/mL | 12 weeks
  The percentage of mothers in each group of pregnant women with HBV DNA below 200,000 IU/mL at the time of delivery will be used as a key secondary efficacy endpoint to evaluate the extent of HBV DNA reduction in mothers receiving TDF/TAF treatment.
The percentage of mothers who experienced HBeAg/HBsAg clearance or seroconversion | 36 weeks
  The percentage of mothers who experienced HBeAg/HBsAg clearance or seroconversion during the study period was used as a secondary efficacy endpoint, and comparisons were made between the two groups.
ALT levels during or after TDF/TAF treatment | 36 weeks
  Observe the proportion of mothers with elevated ALT levels during or after TDF/TAF treatment (i.e., levels 5.1 to 10 times the upper limit of normal) or severe ALT elevation (levels more than 10 times the upper limit of normal), and conduct stratified and subgroup analyses after discontinuation of TDF/TAF (at delivery or at 12 weeks postpartum).
Renal function parameters of pregnant women | 36 weeks
  Summarize the percentage changes in renal function parameters (especially the decline in renal function indicators) of pregnant women in each group during and after antiviral treatment, and analyze the differences between the two groups.
Adverse events (including obstetric complications and laboratory abnormalities) | 36 weeks
  Summarize the percentage of mothers or infants experiencing adverse events (including obstetric complications and laboratory abnormalities) during the comparative study period, and analyze the differences between the two groups.
Proportion of two groups that discontinued treatment due to adverse events | 36 weeks
  Summarize the comparison of the proportion of two groups that discontinued treatment due to adverse events, and evaluate the differences in tolerance and medication adherence to TDF/TAF therapy.
Health-related quality of life (HRQoL) indicators of pregnant women | 36 weeks
  Use the 36-Item Short Form Health Survey (SF-36) to elucidate the differences in quality of life between pregnant women treated with Tenofovir Disoproxil Fumarate (TDF) and those receiving Tenofovir Alafenamide (TAF).The SF-36 scores range from 0 to 100, with higher scores indicating a better quality of life.
Health-related quality of life (HRQoL) indicators of pregnant women | 36 weeks
  Use he Chronic Liver Disease Questionnaire (CLDQ) to elucidate the differences in quality of life between pregnant women treated with Tenofovir Disoproxil Fumarate (TDF) and those receiving Tenofovir Alafenamide (TAF). The CLDQ is scored between 29 and 203, where increased scores reflect improved well-being.
Health-related quality of life (HRQoL) indicators of pregnant women | 36 weeks
  Use Patient Health Questionnaire-9 (PHQ-9) to elucidate the differences in quality of life between pregnant women treated with Tenofovir Disoproxil Fumarate (TDF) and those receiving Tenofovir Alafenamide (TAF). The PHQ-9 is scored from 0 to 27, with lower scores signifying a higher quality of life.

OTHER OUTCOMES:
HBV DNA levels below 20 IU/mL | 12 weeks
  Summarize the percentage difference in HBV DNA levels below 20 IU/mL during delivery between the two groups of pregnant women.
Placental abnormalities | 12 weeks
  Evaluate and compare the percentage of mothers with placental abnormalities in the two groups.
Change in bone mineral density | 36 weeks
  Evaluate the percentage of change (especially decline) in bone mineral density (BMD) among maternal groups during antiviral treatment and after the treatment ends.
Depression, MASLD, or liver fibrosis | 36 weeks
  Evaluate the percentage of mothers with depression, MASLD, or liver fibrosis in each group before using TAF/TDF, during antiviral treatment, and after treatment.

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Guangzhou Eighth People's Hospital, Guangzhou Medical University, Guangzhou, Guangdong
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Shenzhen Baoan Women's and Children's Hospital, Shenzhen, Guangdong
  - Shijiazhuang Maternity & Child Healthcare Hospital, Shijiazhuang, Hebei
  - The Fifth Hospital of Shijiazhuang, Shijiazhuang, Hebei
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing You 'an Hospital, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: Yes
The investigators are committed to the responsible sharing of anonymized Individual Patient Data (IPD) with qualified external researchers upon request or as required by law and/or regulation, based on the following criteria:
  1. Nature of the Request: The specific details and objectives of the data request will be reviewed to ensure alignment with ethical standards and research integrity.
  2. Merit of the Proposed Research: The proposed research's potential scientific value and contribution to the broader scientific community will be evaluated. Priority will be given to research that addresses significant clinical or scientific questions.
  3. Availability of the Data: The feasibility of sharing the requested data, considering any technical, legal, or logistical constraints, will be assessed.
  4. Intended Use of the Data: The intended use of the data will be scrutinized to ensure it is appropriate